CLINICAL TRIAL: NCT01235078
Title: An Observational Study of Intraosseous Vascular Access Compared to Central Venous Catheters in the Emergency Department
Brief Title: Observation of Intraosseous Vascular Access in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Organization: Teleflex (Industry)
Other Study IDs: 2010-04
Record Dates: First submitted 2010-11-03; First posted 2010-11-05 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2012-06

CONDITIONS: Patients Requiring Urgent Vascular Access

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intraosseous vascular access: subjects with urgent vascular access needs in whom intraosseous vascular access has been attempted and/or established.
  Interventions: Device: EZ-IO

INTERVENTIONS:
Device: EZ-IO — powered intraosseous vascular access system
  Other Names: EZ-IO by Vidacare, Powered intraosseous vascular access

SUMMARY:
The purpose of this study is to evaluate the use of powered intraosseous vascular access (EZ-IO by Vidacare) in the emergency department for patients requiring urgent vascular access. Data collected will be compared to historical data on central venous catheter use in the emergency department. The primary hypothesis is that powered intraosseous vascular access will decrease the amount of time needed to obtain vascular access.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring vascular access who would otherwise receive a central venous catheter due to lack of other options.

Exclusion Criteria:

* Fracture in target bone, or significant trauma to the site
* Excessive tissue and/or absence of adequate anatomical landmarks in target bone
* Infection in target area
* IO insertion in past 24 hours, prosthetic limb or joint or other significant orthopedic procedure in target bone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients requiring urgent vascular access
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Time to vascular access | at time of patient's arrival to emergency department, average within 10 minutes
  Time from opening intraosseous device packaging to initial infusion of drugs or fluids via the intraosseous route.

SECONDARY OUTCOMES:
Incidence of complications with intraosseous device | time subject has intraosseous vascular access, an average of 24 hours
  Reported complications by intraosseous device operators.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Gulf Breeze Hospital, Gulf Breeze, Florida
  - Baptist Hospital Pensacola, Pensacola, Florida
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Omaha Children's Hospital and Medical Center, Omaha, Nebraska
  - Methodist Healthcare, University Hospital, Memphis, Tennessee
  - Texas Tech University Medical Center, El Paso, Texas